CLINICAL TRIAL: NCT03830502
Title: Driving Factors of Decision Making for Prophylactic Salpingectomy Versus Tubal Ligation at the Time of Cesarean Section
Status: Completed | Type: Observational
Sponsor: Bartin State Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Yassa, Principal Investigator, Bartin State Hospital
Other Study IDs: EtfalSalp
Record Dates: First submitted 2019-02-03; First posted 2019-02-05 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2020-04

CONDITIONS: Salpingectomy; Sterilization, Tubal
Keywords: Prophylactic salpingectomy; Opportunistic salpingectomy; Risk-reducing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Salpingectomy: Women who gave consent for opportunistic prophylactic bilateral salpingectomy during cesarean section as a Surgical sterilization procedure
  Interventions: Procedure: Surgical sterilization
- Tubal ligation: Women who refused salpingectomy and gave consent for tubal ligation during cesarean section as a Surgical sterilization procedure
  Interventions: Procedure: Surgical sterilization

INTERVENTIONS:
Procedure: Surgical sterilization — Surgical sterilization either standard salpingectomy or tubal ligation with Pomeroy technique

SUMMARY:
Prophylactic (Opportunistic) salpingectomy is a cost-effective strategy recommended for reducing the risk of ovarian cancer at the time of gynecologic surgery in women who have completed childbearing. Similar evidence for cesarean section is growing. However, salpingectomy refers to the surgical removal of a female reproductive organ. Some women may have hesitations about salpingectomy with regard to religious concerns, reduced self-image, tubal reanastomosis or lack of knowledge.

The investigators aimed to explore the underlying factors that motivate women for either decisions.

DETAILED DESCRIPTION:
Prophylactic and opportunistic bilateral salpingectomy is an increasing trend among surgeons and also proven as an effective risk-reducing method for ovarian cancer.

The investigators have experienced denials among women who were seeking tubal ligation as a sterilization procedure during cesarean section after a comprehensive counseling for prophylactic salpingectomy. Therefore, the investigators aimed to assess the driving factors of decision making for prophylactic salpingectomy or tubal ligation. It is planned to preoperatively have a non-validated questionnaire for the women after a detailed briefing.

ELIGIBILITY:
Inclusion Criteria:

* Women seeking for surgical sterilization during their cesarean section
* Elective and Category 2 or more planned cesarean sections

Exclusion Criteria:

* Clinical conditions that lead to planned cesarean hysterectomy such as placenta percreata
* History of ovarian cancer, previous chemotherapy or radiation
* Women who previously underwent sterilization

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who aged over 18 years old and seek for sterilization at the time of cesarean section.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2019-02-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Motivators for sterilization type | Evaluation at preoperative 32th gestational weeks
  A non-validated data collection tool with open-ended questions assessing the factors behind the decision of salpingectomy or tubal ligation. Data collection tool questions why patients choosed or refused salpingectomy in detail. It is not a scale and does not have a range.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, M.D., Principal Investigator — Specialist
Locations (3):
- Turkey (Türkiye) (3):
  - Bartin State Hospital, Bartın
  - Istanbul Sisli Hamidiye Etfal Training And Research Hospital, Health Sciences University, Istanbul
  - Medicalpark Gaziosmanpasa Hospital, Istinye University, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zamorano AS, Mutch DG. Postpartum salpingectomy: a procedure whose time has come. Am J Obstet Gynecol. 2019 Jan;220(1):8-9. doi: 10.1016/j.ajog.2018.09.041. No abstract available. PMID 30591122